CLINICAL TRIAL: NCT00744666
Title: IntraVitreal Triamcinolone Acetonide: Preventing Raised Eye-pressure by Tracking Elevations After Topical Steroids
Acronym: IVTA:PRE-TREAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hotel Dieu Hospital (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr. Kenneth Eng, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 07142008
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Vitreoretinal Disease; Ocular Hypertension
Keywords: Intravitreal triamcinolone acetonide; Side-effects; Ocular hypertension; Glaucoma; Prevention; Vitreoretinal diseases requiring IVTA for treatment
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Prednisolone; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients receive Prednisolone 1% 1gtt qid x 4 weeks. If the intraocular pressure (IOP) after the 4 weeks is > or equal to 21 mmHg, then IVTA will be withheld. If the IOP < 21mmHg, then patients will receive an injection of IVTA.
  Interventions: Drug: Prednisolone 1% topical eye drops
- 2 (No Intervention): Patients will receive an injection of IVTA (no trial of Prednisolone gtts is given).

INTERVENTIONS:
Drug: Prednisolone 1% topical eye drops — Prednisolone 1% 1gtt qid to the eye requiring IVTA
  Arms: 1

SUMMARY:
Intravitreal triamcinolone acetonide (IVTA) is a commonly employed treatment for various vitreoretinal disorders. However, approximately 23% to 50% of patients who receive IVTA develop ocular hypertension after the drug is injected into the eye. Similar to IVTA, topically administered corticosteroids eye drops result in ocular hypertension in approximately 33% of the population. It is unknown whether identifying patients who develop ocular hypertension from topical corticosteroids could be used to identify patients who are at risk for injectable IVTA. Therefore, the purpose of this study is to evaluate the efficacy of topical prednisolone 1% four times daily for one month as a screening test to reduce the incidence and severity of ocular hypertension after IVTA injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with vitreoretinal disease for which IVTA has been chosen as treatment

Exclusion Criteria:

* < 18 years old
* Pregnancy
* Breast feeding
* hx of uveitis
* hx of neovascularization of the iris or anterior chamber angle
* hx of ocular herpes simplex keratitis
* hx of glaucoma
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
To detect a 60% or greater decrease of developing ocular hypertension (>20 mmHg) in the group of patients who received a trial of prednisolone 1% gtts x 4 weeks, compared the group who did not receive a trial of topical prednisolone. | Monthly for 6 months

SECONDARY OUTCOMES:
Visual Acuity | Monthly for 6 months
Incidence of other complications (cataract, retinal detachment, endophthalmitis) | Monthly for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Eng, MD, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre; Jeffery Gale, MD, FRCSC, Principal Investigator — Hotel Dieu Hospital
Locations (4):
- Canada (4):
  - Hotel Dieu Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Jonas JB, Kreissig I, Degenring R. Intraocular pressure after intravitreal injection of triamcinolone acetonide. Br J Ophthalmol. 2003 Jan;87(1):24-7. doi: 10.1136/bjo.87.1.24. PMID 12488256